CLINICAL TRIAL: NCT07067385
Title: Exploratory Clinical Study of Neoantigen Tumor Vaccine Therapy for Gastrointestinal Solid Tumors
Brief Title: Personalized mRNA Cancer Vaccine for Gastrointestinal Solid Tumor Treatment
Acronym: PCV-GSTT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: deepGeneAI (Unknown); Bio-X Institutes, Shanghai Jiao Tong University (Unknown)
Responsible Party: Principal Investigator, Hao Li, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZ202401
Record Dates: First submitted 2025-06-24; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Personalized Neoantigen Vaccine in Combination With Anti-PD-1 Inhibitors in Standard Therapy-Failed and Adjuvant Therapy; Gastrointestinal Tumors
Keywords: neoantigen; p-MHC-TCR; CRC; mRNA; machine learning
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoantigen Personalized Cancer Vaccine (Experimental): Cohort 1: Salvage Therapy ; Cohort 2: Adjuvant Therapy
  Interventions: Biological: Neoantigen Personalized Cancer Vaccine

INTERVENTIONS:
Biological: Neoantigen Personalized Cancer Vaccine — Cohort 1: subjects will receive neoantigen tumor vaccine combination with Sintilimab. Cohort 2: subjects will receive neoantigen tumor vaccine combination with Sintilimab and chemotherapy .
  Other Names: deepGeneAI-001

SUMMARY:
Evaluating the efficacy and safety of Neoantigen Personalized Cancer Vaccine deepGeneAI-001 in combination with Sintilimab in the treatment of Gastrointestinal Solid Tumors

DETAILED DESCRIPTION:
This is a single-center, open, single-arm exploratory clinical study to evaluate the efficacy and safety of Neoantigen Personalized Cancer Vaccine deepGeneAI-001 in combination with Sintilimab in the treatment of Gastrointestinal Solid Tumors, and to provide more clinical treatment options for gastrointestinal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signs the informed consent form, and has good compliance.
2. Male or female, aged 18 years or older.
3. Patients with advanced gastrointestinal tumors: histologically and/or cytologically confirmed recurrent or metastatic gastrointestinal solid tumors not amenable to surgical or local curative treatment, with at least one measurable lesion as defined by RECIST v1.1. Eligible patients must have experienced disease progression following standard antitumor therapy or be unable or unwilling to receive standard treatment.

   Patients with resectable gastrointestinal solid tumors for adjuvant treatment: tumors must be confirmed as completely resected (R0 or R1) by postoperative histopathology, with no prior neoadjuvant therapy, and assessed as fully resectable by imaging.
4. Neoantigen load requirement: at least 10 predicted neoantigen epitopes.
5. The subject must have a tumor lesion suitable for repeated sampling for sequencing and immune testing. Fresh or archived tumor tissue is required, preferably from surgical or core needle biopsy (CNB) samples, including both tumor and 2-3 soybean-sized peritumoral tissues. Paraffin blocks or at least 10-20 unstained tumor tissue sections (4-6 μm thick) with tumor content >20% are acceptable. If the subject cannot provide suitable samples but meets other inclusion/exclusion criteria, the investigator may still consider enrollment.
6. ECOG performance status of 0 or 1.
7. Life expectancy of at least 6 months.
8. Adequate organ and hematologic function, with no severe dysfunction of the heart, lungs, liver, kidneys, or immune system, based on the following laboratory values:

1). Hematology: ANC ≥ 1.5 × 10⁹/L, WBC ≥ 3 × 10⁹/L, PLT ≥ 100 × 10⁹/L, HGB ≥ 90 g/L. Within one week before screening, the subject must not have received blood or platelet transfusions, G-CSF, or erythropoietin (EPO); 2). Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula); 3). Liver function: AST and ALT ≤ 3 × ULN (≤ 5 × ULN for patients with liver cancer or liver metastases); TBIL ≤ 1.5 × ULN (patients with Gilbert's syndrome: TBIL < 3 × ULN); 4). Coagulation: INR ≤ 2 × ULN or APTT ≤ 1.5 × ULN (except for patients on anticoagulants); 5). Endocrine function: TSH within normal limits. Note: If baseline TSH is outside the normal range but free T3 and free T4 are within normal limits, the subject is still eligible.

9. Agrees to provide peripheral blood samples and, optionally, fresh peritumoral tissue for sequencing.

10. Male subjects with reproductive potential and female subjects of childbearing potential agree to use effective contraception from the time of informed consent until 6 months after the last dose of investigational drug.

* Women of childbearing potential include premenopausal women and those within 2 years post-menopause.
* A negative serum pregnancy test is required within 7 days before the first dose of the investigational product.

Exclusion Criteria:

1. Known allergy or hypersensitivity to any investigational drug or its components used in this study.
2. Use of high-dose corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days before the first dose of study drug.
3. Receipt of the following therapies or interventions within 28 days before the first dose of study drug:

   1. Participation in an interventional clinical study;
   2. Major surgery or traumatic injury, or expected to undergo major surgery during the study (minor procedures such as core needle biopsy or placement of a vascular access device within 7 days before the first dose are permitted);
   3. Vaccination with a live attenuated vaccine, or planned vaccination during the study or within 5 months after the last dose of study treatment;
   4. Systemic antitumor therapy (including chemotherapy, small molecule targeted therapy, antibody therapy, cellular immunotherapy, hormonal therapy), or local antitumor therapy (e.g., radiotherapy). Palliative radiotherapy for bone metastases completed >2 weeks before baseline tumor assessment is allowed. Also includes prior treatment with systemic immune-stimulating agents (e.g., interferons or interleukin-2).
4. Presence of severe chronic or active infection within 28 days before the first dose, including but not limited to hospitalization due to infection, sepsis, or severe pneumonia, or any active infection deemed to compromise patient safety by the investigator. Systemic antibiotic treatment within 2 weeks before study start.
5. Clinically significant residual toxicity (≥ grade 2 per CTCAE v5.0) from previous treatment (including systemic therapy, radiotherapy, or surgery), except for alopecia, hyperpigmentation, or other AEs deemed by the investigator not to affect study safety and where recovery to grade ≤1 is not required.
6. Presence of central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may be eligible if neurologically stable for at least 3 months, show no evidence of progression by imaging within 4 weeks before study drug initiation, have recovered from all neurologic symptoms, show no evidence of new or enlarging lesions, and have discontinued corticosteroids, surgery, or radiotherapy for at least 28 days. Carcinomatous meningitis is exclusionary regardless of stability.
7. Active hepatitis B virus (HBV) infection (defined as HBsAg positive and HBV-DNA > 500 IU/mL), hepatitis C virus (HCV) infection (defined as HCV-Ab positive and HCV-RNA positive), human immunodeficiency virus (HIV) infection (HIV-Ab positive), active tuberculosis, or any other active infection requiring systemic treatment within 14 days before first study drug administration (prophylactic anti-infective treatment is allowed).
8. History of clinically significant cardiovascular or cerebrovascular disease within 6 months before the first dose, including but not limited to:

   1. Acute myocardial infarction;
   2. Unstable angina;
   3. Stroke (excluding asymptomatic lacunar infarction not requiring intervention);
   4. History of significant ventricular arrhythmias (e.g., sustained VT, VF, torsades de pointes);
   5. NYHA class III or IV congestive heart failure;
   6. QTcF ≥ 470 ms or history/family history of congenital long QT syndrome;
   7. Baseline left ventricular ejection fraction (LVEF) < 50% or significant wall motion abnormalities on echocardiography;
   8. Poorly controlled hypertension (systolic BP > 160 mmHg or diastolic BP > 100 mmHg);
   9. Other arrhythmias deemed unsuitable by the investigator.
9. Active autoimmune diseases requiring systemic treatment (e.g., corticosteroids or immunosuppressants) within 2 years before the first study dose. Physiologic replacement therapy (e.g., levothyroxine, insulin, or corticosteroids for adrenal or pituitary insufficiency) is permitted.
10. History of other malignancies within 3 years before study treatment, except for those with curative potential after radical treatment, such as basal or squamous cell skin cancers, localized low-risk prostate cancer, papillary thyroid carcinoma, or any in situ carcinoma (e.g., cervical carcinoma in situ or ductal carcinoma in situ).
11. Any other severe or uncontrolled disease or condition that, in the opinion of the investigator, could interfere with study participation or compliance, including but not limited to:

    1. Severe respiratory disease, such as interstitial lung disease, severe asthma, idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or evidence of active pneumonia on screening chest CT;
    2. Severe venous or arterial thromboembolism, such as pulmonary embolism or deep vein thrombosis (excluding asymptomatic, untreated intermuscular venous thrombosis);
    3. Symptomatic or large pleural effusion or ascites requiring symptomatic management;
    4. Active or past history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis);
    5. Symptomatic or significant pericardial, pleural, or abdominal effusion on screening;
    6. Tumors encasing major blood vessels or with extensive necrosis or cavitation on imaging, which the investigator considers to pose a bleeding risk;
    7. History of gastrointestinal perforation, surgical/wound healing complications, or significant bleeding events.
12. Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
13. History of substance abuse or psychiatric disorder that may interfere with compliance.
14. Pregnant or breastfeeding women. Pregnancy is defined as the period from conception until the end of gestation. Pregnancy status must be confirmed by a serum hCG test within 7 days before study initiation.
15. Prior treatment with cell therapies (e.g., TCR-T, CAR-T, TILs) or neoantigen-based cancer vaccines. Prior treatment with immune checkpoint inhibitors (e.g., PD-1, PD-L1). Receipt of immune-stimulating agents (e.g., thymosin, interferon, interleukin-2) within 6 weeks before study treatment.
16. Genetic sequencing reveals functional defects in genes related to antigen presentation, antigen recognition, or cytotoxicity.
17. Any other condition deemed inappropriate for study enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events as graded by CTCAE v5.0 | Up to 2.5 years
Serious adverse events as graded by CTCAE v5.0 | Up to 2.5 years
Immunogenicity of a personalized cancer vaccine as measured by interferon-γ secreting T lymphocytes in peripheral blood mononuclear cells (PBMCs) using ELISpot | Up to 2.5 years

SECONDARY OUTCOMES:
Cohort 1: Objective Response Rate (ORR) by RECIST 1.1 | Up to 2.5 years
Cohort 1: Duration of Response (DOR) | Up to 2.5 years
Cohort 1: Disease Control Rate (DCR) | Up to 2.5 years
Cohort 1: Progression Free Survival (PFS) as assessed by RECIST 1.1 | Up to 2.5 years
Cohort 1: Overall Survival (OS) | Up to 2.5 years
Cohort 2: 18-month Recurrence-free survival (RFS) rate | Up to 2.5 years
Cohort 2: 18-month Overall Survival (OS) rate | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hao Li, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, SH, China

IPD SHARING:
Plan to Share IPD: No
The investigators decide not to share.